CLINICAL TRIAL: NCT00912405
Title: A Clinical Evaluation of the Steroid-Eluting Sinexus Intranasal Splint When Used Following Functional Endoscopic Sinus Surgery in Patients With Chronic Sinusitis
Brief Title: Clinical Evaluation of the Steroid-Eluting Sinexus Intranasal Splint When Used Following Functional Endoscopic Sinus Surgery (FESS) in Patients With Chronic Sinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P500-0209
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Sinusitis
Keywords: Patients diagnosed with Chronic Sinusitis undergoing functional endoscopic surgery (FESS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sinexus Intranasal Splint (Experimental): Patient receives a drug-coated intranasal splint
  Interventions: Device: Steroid-Eluting Sinexus Intranasal Splint

INTERVENTIONS:
Device: Steroid-Eluting Sinexus Intranasal Splint — Intranasal drug-coated splint placed after functional endoscopic surgery (FESS)

SUMMARY:
This study allows continued access to the Sinexus Intranasal Splint while a marketing application is being prepared. This study will generate additional performance, reimbursement and safety data for the steroid-eluting Sinexus Intranasal Splint when used following Functional Endoscopic Sinus Surgery (FESS) in patients with chronic sinusitis (CS).

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has a diagnosis of chronic sinusitis
* Patient has a clinical indication for and has consented to FESS
* Patient CT scan confirms CS diagnosis within 6 months of procedure
* CT sacn confirms presence of disease in ethmoid sinus(es)
* Planned FESS includes unilateral or bilateral total ethmoidectomy

Exclusion Criteria:

* Immune deficiency (IGG subclass deficiency or IGA deficiency)
* Oral-steroid dependent COPD, asthma or other condition
* Clinical evidence of acute bacterial sinusitis
* History or diagnosis of glaucoma or ocular hypertension
* Clinical evidence or suspicion of invasive fungal sinusitis
* Evidence of disease or condition expected to compromise survival or ability to complete follow-up
* Known history of allergy or intolerance to corticosteroids
* History of insulin dependent diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Central California Ear, Nose Thraot, Fresno, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sinexus Intranasal Splint
Started | 50
Completed | 45
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Sinexus Intranasal Splint
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 50
Lund MacKay CT Stage [Mean (Standard Deviation); unit: units on a scale] — The Lund Mackay CT Staging system is a scale ranging from 0 to 24, where lower scores represent a better condition. each sinus is scored 0, 1 or 2, where 0=no opacification, 1=partial opacification and 2=complete opacification. 12 areas of the anatomy are evaluated, resulting in the scale ranging from 0 to 24.
  units on a scale | 11.2 (5.5)
Proportion of Patients with Polyps [Number; unit: participants] | 33
Proportion of Patients Undergoing Revision Surgery [Number; unit: participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety as Determined by the Frequency of Serious Adverse Local Tissue Response (SALT)
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: Number of Sinuses
Units Other Than Participants: number of sinuses
Arm/Group | Sinexus Intranasal Splint
Number analyzed (Participants) | 50
Number analyzed (number of sinuses) | 90
Number of Sinuses | 6 [2.49 to 13.95]

2. Primary Outcome: Device Placement Success Rate
Description: A proportion where the numerator is the number of successful device placements and denominator is the number of attempted sinuses.
Time Frame: At the time of procedure
Measure: Number; unit: Sinuses
Units Other Than Participants: Sinuses Attempted
Arm/Group | Sinexus Intranasal Splint
Number analyzed (Participants) | 50
Number analyzed (Sinuses Attempted) | 90
Sinuses | 90

3. Secondary Outcome: Assessment of Changes From Baseline in Intra-ocular Pressure and Lens Opacities
Description: Ocular safety was characterized by assessing the frequency and severity of changes from baseline in intra-ocular pressure and lens opacities. No specific pass/fail criteria we specified.
Time Frame: Baseline and 30 days
Measure: Number; unit: Pts. w/ significant IOP elevation
Arm/Group | Sinexus Intranasal Splint
Number analyzed (Participants) | 50
Pts. w/ significant IOP elevation | 0

4. Secondary Outcome: Number of Sinuses With Significant Post-operative Adhesion Formation
Description: Adhesions were graded on a 5 point categorical scale with grades 3 and 4 considered clinically significant. 0=none, 1=small/non-obstructing, 2=obstructing/easily separated, 3=dense/obstructing/difficult to separate, and 4=severe/complete adhesion to lateral nasal wall.
Time Frame: 30 days
Measure: Number; unit: sinuses
Units Other Than Participants: Sinuses
Arm/Group | Sinexus Intranasal Splint
Number analyzed (Participants) | 50
Number analyzed (Sinuses) | 90
sinuses | 1

ADVERSE EVENTS:
Arm/Group | Sinexus Intranasal Splint
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 23/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sinexus Intranasal Splint (N=50)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sinexus Intranasal Splint (N=50)
Headache (General disorders) | 5 (5)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No